CLINICAL TRIAL: NCT06990438
Title: Effect of Long-Term Use of Tenofovir (TDF) on Bone Density in Patients With Chronic Hepatitis B
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nour shaaban Mohamed Abd elrasoul, Principal Investigator, Assiut University
Other Study IDs: TDF ON BONE HEALTH
Record Dates: First submitted 2025-05-17; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Tenofovir Disoproxil Fumarate; Bone Density; Chronic HBV Infection
MeSH Terms: interventions — Tenofovir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: TDF (Tenofovir) — ANTIVIRAL TREATMENT FOR CHRONIC HEPATITIS B VIRUS INFECTION

SUMMARY:
This study aims to evaluate the effect of long-term use of Tenofovir Disoproxil Fumarate (TDF) on bone density in patients with chronic hepatitis B virus (HBV) infection. Tenofovir is a widely used antiviral medication for the treatment of HBV. While it is generally well tolerated, some studies have reported potential adverse effects on bone mineral density, particularly with long-term use.

The objective of this research is to assess whether extended TDF therapy is associated with reduced bone density or increased risk of osteopenia or osteoporosis in adult patients with chronic HBV infection. The study will involve clinical evaluation and radiological assessment of bone health using dual-energy X-ray absorptiometry (DEXA) scans, as well as relevant biochemical markers.

This investigation will provide important data on the long-term safety profile of Tenofovir in relation to bone health and help guide future clinical decisions for the management of chronic hepatitis B.

DETAILED DESCRIPTION:
Hepatitis B is a viral infection that affects approximately 257 million people worldwide, with an estimated 820,000 deaths annually due to HBV-related complications. It is a leading cause of liver cirrhosis and hepato-cellular carcinoma (HCC), making it a major global public health concern .

The diagnosis of Chronic Hepatitis B (CHB) is established by the persistence of Hepatitis B surface antigen (HBsAg) for more than six months . Some patients with chronic HBV infection may experience acute exacerbation, potentially progressing to acute-on-chronic liver failure (ACLF), a condition with a high mortality rate despite intensive supportive care and resource utilization. While liver transplantation is considered a potential life-saving treatment for ACLF, its widespread clinical application is limited due to donor shortages and high financial costs. Therefore, early intervention and treatment are crucial in managing patients with ACLF .

The primary goals of antiviral therapy in CHB are to suppress viral replication and promote the loss of HBV-related antigens . Currently, there are two major classes of antiviral agents approved for treating CHB: Interferon-Alpha and Nucleos(t)ide Analogues (NUCs). Among the NUCs, Entecavir (ETV), Tenofovir Disoproxil Fumarate (TDF), and Tenofovir Alafenamide (TAF) are the most widely used first-line treatments. These agents are effective, orally administered, and generally well-tolerated. However, long-term treatment is often required, as premature discontinuation may lead to virological relapse and liver failure.

TDF is considered one of the most potent antiviral agents against both HBV and HIV. However, it has been associated with bone toxicity, primarily through the development of osteoporosis via multiple mechanisms. Intracellular accumulation of TDF can lead to proximal tubular dysfunction and Fanconi syndrome, resulting in hypophosphatemic osteomalacia . Additionally, TDF has been shown to reduce osteoblast gene expression, impairing osteoblast function and decreasing bone formation .

Moreover, TDF-induced reduction in phosphate reabsorption in the proximal renal tubules can lead to bone disease, including hypouricemia and hypophosphatemia, ultimately contributing to osteomalacia and an increased risk of fractures. In contrast, TAF exhibits greater plasma stability, and therefore, its impact on renal and bone toxicity may be significantly lower

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

Adult male or female patients aged 18 to 60 years.

Diagnosed as HBV-positive.

Long-term use of Tenofovir Disoproxil Fumarate (TDF) for more than five years.

Exclusion Criteria:

Presence of other chronic liver diseases.

Diagnosed with Chronic Kidney Disease (CKD), regardless of etiology.

Patients who refuse to participate in the study.

Patients on combination therapy, including:

Interferon and Nucleoside analogue combination therapy.

Multiple nucleoside analogue combination therapy.

-

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study Population Age Range: 18 to 60 years Sex: Male and Female HBV Status: HBV-positive patients Treatment Duration: Long-term use of Tenofovir (TDF) for more than five years Sampling Method: Non-Probability Sampling Healthy Volunteers: Not Accepted
Sampling Method: Non-Probability Sample
Enrollment: 172 (Estimated)
Dates: Start 2025-05-22 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Bone Mineral Density (BMD) | Baseline to 5 years post-TDF initiation
  Change in BMD measured by dual-energy X-ray absorptiometry (DEXA), expressed as percentage change from baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Assuit, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Han Y, Zeng A, Liao H, Liu Y, Chen Y, Ding H. The efficacy and safety comparison between tenofovir and entecavir in treatment of chronic hepatitis B and HBV related cirrhosis: A systematic review and Meta-analysis. Int Immunopharmacol. 2017 Jan;42:168-175. doi: 10.1016/j.intimp.2016.11.022. Epub 2016 Dec 1. PMID 27915131
- [Result] Kara AV, Yildirim Y, Ozcicek F, Aldemir MN, Arslan Y, Bayan K, Celen MK. Effects of entecavir, tenofovir and telbivudine treatment on renal functions in chronic hepatitis B patients. Acta Gastroenterol Belg. 2019 Apr-Jun;82(2):273-277. PMID 31314188
- [Result] Perazella MA. Tenofovir-induced kidney disease: an acquired renal tubular mitochondriopathy. Kidney Int. 2010 Dec;78(11):1060-3. doi: 10.1038/ki.2010.344. PMID 21076445
- [Result] Jeong S, Shin HP, Kim HI. Real-World Single-Center Comparison of the Safety and Efficacy of Entecavir, Tenofovir Disoproxil Fumarate, and Tenofovir Alafenamide in Patients with Chronic Hepatitis B. Intervirology. 2022;65(2):94-103. doi: 10.1159/000519440. Epub 2021 Nov 3. PMID 34731856
- [Result] Trepo C, Chan HL, Lok A. Hepatitis B virus infection. Lancet. 2014 Dec 6;384(9959):2053-63. doi: 10.1016/S0140-6736(14)60220-8. Epub 2014 Jun 18. PMID 24954675
- [Result] Nguyen MH, Wong G, Gane E, Kao JH, Dusheiko G. Hepatitis B Virus: Advances in Prevention, Diagnosis, and Therapy. Clin Microbiol Rev. 2020 Feb 26;33(2):e00046-19. doi: 10.1128/CMR.00046-19. Print 2020 Mar 18. PMID 32102898
- [Result] Chien RN, Liaw YF. Current Trend in Antiviral Therapy for Chronic Hepatitis B. Viruses. 2022 Feb 21;14(2):434. doi: 10.3390/v14020434. PMID 35216027
- [Result] Castillo AB, Tarantal AF, Watnik MR, Martin RB. Tenofovir treatment at 30 mg/kg/day can inhibit cortical bone mineralization in growing rhesus monkeys (Macaca mulatta). J Orthop Res. 2002 Nov;20(6):1185-9. doi: 10.1016/S0736-0266(02)00074-8. PMID 12472227
- [Result] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Result] Terrault NA, Bzowej NH, Chang KM, Hwang JP, Jonas MM, Murad MH; American Association for the Study of Liver Diseases. AASLD guidelines for treatment of chronic hepatitis B. Hepatology. 2016 Jan;63(1):261-83. doi: 10.1002/hep.28156. Epub 2015 Nov 13. No abstract available. PMID 26566064